CLINICAL TRIAL: NCT02588066
Title: Pancreatoduodenectomy With or Without Prophylactic Ligamentum Teres Hepatic Wrap Around the Gastroduodenal Artery Stump for Prevention of Pancreatic Hemorrhage - Panda - Multicentric Randomized Controlled Trial
Brief Title: Pancreatoduodenectomy With or Without Ligamentum Teres Wrap Around Gastroduodenal Artery Stump for Prevention of Pancreatic Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TW-002
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Pancreatoduodenectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Index test (Experimental): Ligamentum teres/falciform-plasty around the gastroduodenal artery stump during pancreatoduodenectomy
  Interventions: Procedure: Ligamentum teres/falciform-plasty
- Reference test (No Intervention): No Ligamentum teres/falciform-plasty around the gastroduodenal artery stump during pancreatoduodenectomy

INTERVENTIONS:
Procedure: Ligamentum teres/falciform-plasty — Ligamentum teres/falciform-plasty around the gastroduodenal artery stump during pancreatoduodenectomy
  Arms: Index test

SUMMARY:
To investigate, whether a prophylactic wrapping of the gastroduodenal artery stump with the ligamentum teres or falciform hepatic (embryological structures, covered with peritoneum that do not have relevant meaning for adults) can reduce the incidence of arrosion bleeding during surgery.

Thus a surgical technique is evaluated prospectively.

DETAILED DESCRIPTION:
Pancreatoduodenectomy is a standard surgical procedure for resection of tumors of the pancreatic head and neck, and for selected patients with chronic pancreatitis. A postoperative pancreatic fistula (POPF) is a severe and frequent complication that may lead to a potentially letal arrosion hemorrhage from the stump of the gastroduodenal artery (GDA). Aim of the study is to evaluate the prophylactic wrapping of the GDA stump using the falciform hepatic ligament during the index operation. The null hypothesis is that prophylactic wrapping does not decrease the incidence of arrosion hemorrhage from the GDA stump. The study is designed as a randomized, single-blinded, controlled, multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective open pancreatoduodenectomy (pylorus-preserving or classic) with pancreatojejunostomy for tumors, or cystic lesions of the pancreatic head, tumors of the distal bile duct, duodenum or for chronic pancreatitis
* american society of anesthesiologists classification I-III
* age ≥18 years
* given informed consent

Exclusion Criteria:

* status post previous abdominal surgery with resection of the falciform ligament (e.g. hemihepatectomy)
* No reconstruction using a pancreatojejunostomy (e.g. pancreatogastrostomy)
* simultaneous visceral arterial resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-11; Primary Completion 2020-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Incidence of arrosion bleeding | >24 hours after partial pancreatoduodenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Welsch, Principal Investigator — Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Germany
Locations (1):
- Department of Surgery, University Hospital Dresden, Dresden, Germany

REFERENCES:
- [Derived] Welsch T, Mussle B, Korn S, Sturm D, Bork U, Distler M, Grahlert X, Klimova A, Trebesius N, Kleespies A, Kees S, Beckert S, Reim D, Friess H, Elwerr M, Kleeff J, Popescu O, Schmitz-Winnenthal H, Janot-Matuschek M, Uhl W, Weber GF, Brunner M, Golcher H, Grutzmann R, Weitz J. Pancreatoduodenectomy with or without prophylactic falciform ligament wrap around the hepatic artery for prevention of postpancreatectomy haemorrhage: randomized clinical trial (PANDA trial). Br J Surg. 2021 Dec 17;109(1):37-45. doi: 10.1093/bjs/znab363. PMID 34746958
- [Derived] Mussle B, Zuhlke L, Wierick A, Sturm D, Grahlert X, Distler M, Rahbari NN, Weitz J, Welsch T. Pancreatoduodenectomy with or without prophylactic falciform ligament wrap around the gastroduodenal artery stump for prevention of pancreatectomy hemorrhage. Trials. 2018 Apr 12;19(1):222. doi: 10.1186/s13063-018-2580-0. PMID 29650056